CLINICAL TRIAL: NCT03572543
Title: Enhancement of Therapeutic Learning in Obsessive-compulsive Disorder Using Transcranial Direct Current Stimulation
Brief Title: Enhancement of Therapeutic Learning in OCD Using tDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1412015006_a; 1K23MH111977 (NIH)
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator): Current will be ramped in/out for 30 seconds at the begging and end of a 20-minute period and a constant current will be delivered for the 20-minutes between ramping.
  Interventions: Device: tDCS
- Sham tDCS (Sham Comparator): Current will be ramped in/out for 30 seconds at the begging and end of a 20-minute period during which no stimulation will be delivered.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Subjects will receive 20 minutes of multifocal transcranial direct current stimulation. The anode will be placed over the frontal pole (Fpz, 10-20 EEG) and will be surrounded by 5 return electrodes (cathodes). Current will be set at 1.5mA and will be ramped in/out at the begging and end of the 20-minutes of stimulation over the course of 30 seconds.
  Other Names: transcranial direct current stimulation; transcranial electrical stimulation; Starstim®

SUMMARY:
Psychiatric disorders characterized by pathological fear and anxiety are common and often disabling. Despite their limitations, exposure therapies are among the most efficacious treatments for these disorders. Extinction learning is thought to be a core mechanism of therapeutic exposure. Extinction learning is mediated by a well-defined circuit encompassing the medial prefrontal cortex (mPFC), amygdala, and hippocampus. This raises the exciting possibility that direct engagement of this circuitry might enhance the response to therapeutic exposure. Transcranial direct current stimulation (tDCS) is a neuromodulation technology that can augment brain plasticity, learning, and memory. The proposed study will evaluate whether tDCS can improve therapeutic learning and memory processes among participants diagnosed with obsessive-compulsive disorder (OCD) This study aims to use tDCS to improve learning and memory processes within the context of an exposure laboratory challenge. Participants diagnosed with OCD will complete a two-day experimental study. On day 1, participants will receive sham (placebo) or active tDCS followed by approximately 50-minutes of individualized exposure. on day 2, participants will return to complete an additional 50-minutes of exposure. Subjective distress will be repeatedly monitored during exposure to allow for the modeling of within-trail and within-session learning and between-session recall of learning.

DETAILED DESCRIPTION:
Most effective behavioral treatments of disordered anxiety involve repeated exposure to feared stimuli, which often results in systematic reductions in fearful responding to said stimuli. It is believed that this process results from successful fear extinction, a well-characterized learning process that is mediated by fear extinction brain circuitry. Namely, fear extinction is an inhibitory learning process that requires activation and plasticity within a variety of brain regions, including the medial prefrontal cortex (mPFC), which can exert inhibitory control over fearful responding and parts of the brain that drive said responding. Behavioral treatments of disordered anxiety, while effective, have serious limitations; many patients fail to respond at all or only partially respond to exposure-based treatments. One candidate reason for this is deficits in fear extinction learning or memory processes. The proposed study aims to examine the effects of non-invasive neuromodulation - namely, multifocal transcranial direct current stimulation (tDCS) targeting the mPFC - on therapeutic learning and memory among adults diagnosed with obsessive-compulsive disorder (OCD).

This study will recruit 26 subjects with OCD to complete a two-day experimental protocol to examine the effects of tDCS on therapeutic learning and memory, which will be measured with an exposure and response prevention laboratory challenge. On Day 1, OCD subjects will be randomized (1:1, double-blind) to receive Active (n = 13) or Sham (n = 13) tDCS prior to completing five 10-minute in vivo exposure exercises to assess the effects of tDCS on the acquisition of therapeutic learning. Subjects and raters (including those directing exposure sessions) will be blind to allocation. On Day 2, OCD subjects will return to complete five additional exposure trials to examine the effects of tDCS on recall of therapeutic learning. Subjective ratings of emotional distress (0-100) will be collected at baseline, before and after tDCS, and during each minute of each exposure trial. It is hypothesized that tDCS will improve the acquisition and recall of therapeutic learning (Aim 4); that participants randomized to Active tDCS would show more rapid reductions in subjective distress and would recall therapeutic learning on Day 2 when compared to participants randomized that Sham tDCS.

tDCS will be delivered using an 8-channel Starstim transcranial electric stimulator from Neuroelectrics. To target the mPFC, the anodal electrode will be placed over the frontal pole (Fpz, 10-20 EEG landmarks) and will be surrounded by five return (cathodal) electrodes in a circumferential array (AF7, AF8, F3, Fz, and F4). Subjects in the Active tDCS condition will receive 20 minutes of direct current stimulation for 20 minutes; current will be ramped in and out for 30 seconds at the beginning and end of the 20-minute period. Subjects in the Sham tDCS condition will receive the same electrode placement and ramping procedures, but no current will be delivered between ramping.

Linear mixed modeling will be used to assess within and between-trial exposure-relevant learning. Power analyses suggest that a sample of 24 (12 per condition) would adequately power a priori analyses when using linear mixed modeling. Mixed ANOVA will be used to assess recall of exposure-relevant learning. The proposed study will provide important preliminary data to examine the potential for medial prefrontal tDCS to augment exposure-relevant therapeutic learning.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent (as established by clinical interview), and voluntary, signed informed consent prior to the performance of any study-specific procedures;
* Ability and willingness to perform study-relevant clinical assessments and tDCS;
* Age 18-55;
* Medication free or stable (> 4 weeks) medication(s).
* A Diagnostic and Statistical Manual diagnosis of OCD; and
* Clinically significant obsessions and compulsions of at least moderate severity, as established by a score of at least 16 on the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) during initial screening.

Exclusion Criteria:

* Any unstable medical, psychiatric, or neurological condition (including active or otherwise problematic suicidality) that may necessitate urgent treatment;
* Any substance dependence or severe substance abuse within the past 6 months;
* Daily use of psychotropic medications that substantially lower seizure threshold (e.g., clozapine);
* Daily use of psychotropic drugs that may interfere with extinction learning (e.g., anxiolytics);
* Any history of a psychotic disorder or of mania;
* Current active suicidal ideation or any suicidal intent;
* Any major neurological disease or history of major head trauma, including concussion with extended loss of consciousness, or of psychosurgery;
* Any history of epilepsy;
* Pregnancy;
* Any metal in the body or other contraindication to MRI scanning or tDCS;
* Any history of adverse effects to brain stimulation;
* Recent (< 8 weeks) change in psychotherapy - i.e. no recently instituted cognitive behavioral therapy will be permitted, but ongoing therapy of long duration will not constitute an exclusion;
* OCD symptoms that cannot be provoked with in vivo exposures in a laboratory environment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2017-09-07 (Actual)

PRIMARY OUTCOMES:
Subjective Units of Distress | Collected every minute up through 50 minutes
  0-100 subjective distress self-report rating

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Adams, PhD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers upon request and review by the PI and relevant collaborators. Data will be stored on a yet to be determined data sharing repository supported by the National Institutes of Health.
Supporting Information: SAP, Analytic Code
Time Frame: Data will be made available following study publication.

REFERENCES:
- [Derived] Adams TG, Cisler JM, Kelmendi B, George JR, Kichuk SA, Averill CL, Anticevic A, Abdallah CG, Pittenger C. Transcranial direct current stimulation targeting the medial prefrontal cortex modulates functional connectivity and enhances safety learning in obsessive-compulsive disorder: Results from two pilot studies. Depress Anxiety. 2022 Jan;39(1):37-48. doi: 10.1002/da.23212. Epub 2021 Aug 31. PMID 34464485